CLINICAL TRIAL: NCT06576492
Title: Assessment of the Effects and Tolerance of the RV4986A Lotion in Men With AGA After Hair Transplant: Controlled and Randomized Open Study
Brief Title: Assessment of the Effects and Tolerance of the RV4986A Lotion in Men With AGA After Hair Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV4986A20200299
Record Dates: First submitted 2024-07-31; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Experimental): Application of RV4986A lotion associated with RD0057H shampoo (Extra Doux shampoo)
  Interventions: Other: RV4986A lotion; Other: RD0057H shampoo
- Control group (Other): Application of RD0057H shampoo (Extra Doux shampoo)
  Interventions: Other: RD0057H shampoo

INTERVENTIONS:
Other: RV4986A lotion — * Application between Month -0.5 and Month 0 (before hair transplant): once a day on the entire scalp
  * From 4 days after hair transplant and until Visit 4 (Month 0,5 post transplant): once a day on the recipient area
  * Between Month 0.5 and Month 12: once a day on the entire scalp
  Arms: Treated group
Other: RD0057H shampoo — * Application between Month -0.5 and Month 0 (before hair transplant): at usual frequency when required on the entire scalp
  * From 2nd day after hair transplant and until the 7th day after hair transplant: application on the recipient area with a spray containing mixture of water and shampoo. For the rest of the head application with the same modalities than before hair transplant
  * From the 8th day after hair transplant to the 15th day: application with a sponge on the recipient area
  * From the 16th day after hair transplant and for the next 12th months: application with the same modalities than before hair transplant

SUMMARY:
Alopecia involves a diminution of visible hair that can have significant psychosocial effects and impairment of quality of life. There are numerous types of alopecia, among them, androgenic alopecia (AGA) is the most common form surgically treatable.

Androgenic alopecia is characterized by progressive visible thinning of scalp hair in genetically susceptible men (MAGA, or male pattern androgenic alopecia) and in some women (FPHL, or female pattern hair loss).

Among the plethora of products available proposed to promote hair growth in the scalp, only 2 medications are approved by the US Food and Drug Administration (FDA). These medications are finasteride (systemic) and minoxidil (topical).

In some cases, limited perceived efficacy of these treatments, poor tolerance, fear and lack of information on treatment duration and possible adverse events may lead to premature stop of treatment, disappointment and influence on patient compliance.

When conventional treatments have proven to be deceptive, a surgical treatment can be considered: hair transplant, that has evolved mainly with the aim of making the results look more and more natural.

Hair transplant, although performed on an outpatient basis, is an invasive technique, with the following immediate side effects: pain, pruritus, inflammation, scabs, swollen eyelids with tearing which last about 15 days. A social exclusion for 15 days after the transplant is generally necessary. For 1 to 2 months, the Red Scalp syndrome or inflammatory scalp is observed.

The growth of transplanted hair starts from the 6th month and the expected result is not really achieved until one year.

The product RV4986A is a non-rinsed cosmetic lotion intended to be used every day on the entire scalp especially in case of hormonal or hereditary chronic hair loss (as AGA) and also before hair transplant in order to prepare hair scalp and after hair transplant in order to soothe the scalp.

To date, no consensus and guidelines for pre- and post-transplant management exist regarding cosmetic products to apply that could limit their transplant side effects in time and intensity.

The aim of the study is to assess the effect of a new product (topical lotion) developed as an adjuvant product pre- and post-transplant that prepares hair scalp before the transplant and soothes it after hair transplant.

ELIGIBILITY:
Main inclusion criteria:

* Male
* Subject requiring hair transplant with micrografts (strip technique or FUE technique)
* Subject aged ≥ 18 years old
* Subject having androgenetic alopecia selected by the investigator for a hair transplant

Main non-inclusion criteria:

* Subject having any other hair disorder or hair disease (telogen effluvium, alopecia areata, cicatricial alopecia, hair shaft disorder, trichotillomania…) and liable to interfere with the study assessments
* Subject having dermatological pathology or evolutive skin lesion on the scalp (psoriasis, seborrheic dermatitis, severe erythema, severe excoriation, severe sunburn, …)
* Iron deficiency (confirmation by ferritin assay results from less than 3 months performed during preoperative assessment)
* Thyroid disorders (confirmation by thyroid hormon assay results from less than 3 months performed during preoperative assessment)
* Systemic treatment with antithyroid or iron supplement established or modified within 3 months before the inclusion or planned during the study
* Radiotherapy or chemotherapy at any time before the inclusion or planned during the study
* Systemic anti-hair loss treatment (anti-androgenic treatments…) established or modified within 6 months before the inclusion visit or planned during the study
* Topical anti-hair loss treatment (Minoxidil…) established or modified within 3 months before the inclusion visit or planned during the study
* Any other systemic treatment (cardiovascular, endocrine, antidepressant, antipsychotic, …) established or modified during the previous weeks before the inclusion or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the products according to the investigator's assessment
* Any other topical treatment or product applied on the scalp within previous weeks before the inclusion or planned during the study that can limit the effectiveness of the transplant and liable to interfere with the study assessments, according to the investigator's opinion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by global aspect of the scalp | Months 0.5, 1, 3, 6, 9 and 12 compared to Month 0 (hair transplant)
  assessed in vivo by the investigator, on the recipient area (frontal and/or vertex areas) on 5-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by hair growth | Months 6, 9, 12 compared to Month 0 (hair transplant)
  assessed in vivo by the investigator, on the recipient area on 5-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by aspect of the scalp | Months 0, 0.5, 6, 9, 12 compared to Month -0.5 (inclusion, pre-hair transplant)
  assessed from standardised photographs, rated by several investigators (or trained people) on blinded groups, on the recipient area on 11-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by aspect of the hair | Months 0, 0.5, 6, 9, 12 compared to Month -0.5 (inclusion, pre-hair transplant)
  assessed from standardised photographs, rated by several investigators (or trained people) on blinded groups, on the recipient area on 11-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Scalp soothing and cosmetic recovery (erythema and scalp oedema evaluation) | Months 0 and 0.5
  Physical signs erythema and scalp oedema scoring (in vivo assessments of) on 11-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Scalp soothing and cosmetic recovery (crusts and healing evaluation) | Months 0, 0.5, 1 and 3
  Physical signs crusts and healing scoring (in vivo assessments of) on 11-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Scalp soothing and cosmetic recovery | Months 0 and 0.5
  Visual evaluation by Trichoscopy of crusts and erythema
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Global efficacy (PGA = patient global assessment) | Months 0, 0.5, 1, 3, 6, 9 and 12 and monthly between each visit
  assessed by the subject on the recipient area, according to a 5-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Functional signs | At each visit from Month 0 (hair transplant)
  assessed by the subject on the recipient area, according to a 11-point scale
Evaluate the effects of the RV4986A lotion on hair and scalp for the first 12 months after hair transplant compared to a control group by Satisfaction & Cosmetic acceptability & Quality of Life & Hair/Scalp perception assessments | Months 0, 1, 6 and 12
  assessed by the subject with subject's questionnaire
Evaluate the tolerance of the products for 12 months of use by adverse events | At each visit from Month 0 to Month 12
  Adverse events
Evaluate the tolerance of the products for 12 months of use by physical and functional signs | At each visit from Month 0 to Month 12
  assessed by the investigator for physical signs and by the subject for functional signs on the entire scalp (before hair transplant) or recipient area (after hair transplant), according to a 11-point scale
Evaluate the tolerance of the products for 12 months of use by global tolerance per subject | at Month 0 (for period of pre-transplant) and at Month 12 (end of the study)
  assessed by the investigator for both groups and per subject, considering all individual AE and their characteristics, based on a 5-point scale
Evaluate the subject's compliance regarding the test product | At each visit from Month 0 to Month 12
  The subject will report his compliance in a subject's diary.
  Compliance will be monitored by weighing tubes. Test products will be weighed at the beginning and the end of the study under sponsor responsibility according a validated weighing protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Medico Ricart, Madrid, Chamartin, Spain

IPD SHARING:
Plan to Share IPD: No